CLINICAL TRIAL: NCT01518946
Title: A Phase 4, Randomized, Double-blind, Placebo-controlled, Crossover Study to Investigate the Clinical Benefit of Midodrine Hydrochloride in Male and Female Subjects With Symptomatic Orthostatic Hypotension
Brief Title: Tilt-Table Study of the Clinical Efficacy of Midodrine in Symptomatic Orthostatic Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD426-406
Record Dates: First submitted 2012-01-18; First posted 2012-01-26 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Orthostatic Hypotension
Keywords: Symptomatic Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midodrine HCl (Active Comparator)
  Interventions: Drug: Midodrine HCl
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midodrine HCl — dose at the subject's current dose level
  Other Names: ProAmatine®
  Arms: Midodrine HCl
Drug: Placebo — single dose of matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether midodrine works against the symptoms of orthostatic hypotension caused by being on a tilt table.

DETAILED DESCRIPTION:
The efficacy of midodrine will be assessed in those subjects who have severe symptoms of orthostatic hypotension when not taking midodrine and are controlled when taking midodrine. The study will involve approximately 4 overnight stays.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects must be 18 years of age or older and ambulatory.
2. Females of child-bearing potential (FOCP) must have a negative serum beta human chorionic gonadotropin (HCG) pregnancy test.
3. A documented history of severe Symptomatic Orthostatic Hypotension (SOH) that, in the judgment of the treating physician, has required treatment with midodrine HCl , and has been at a stable dose for at least 3 months.
4. The subject has manifested at least 1 of the following symptoms while standing or had a medical history of 1 of the following when not treated for orthostatic hypotension (OH): dizziness, lightheadedness, feeling faint, or feeling like they might black out.

Exclusion Criteria:

1. The subject is a pregnant or lactating female.
2. The subject has pre-existing sustained supine hypertension greater than 180mmHg systolic and 110mmHg diastolic BP or had these measurements at the Screening Visit. Sustained is defined as persistently greater at 2 separate measurements at least 5 minutes apart with the subject supine and at rest for the 5 minutes.
3. Subjects taking concomitant medications of interest are excluded unless those medications are reviewed and discussed with the Medical Monitor or Study Physician and documented prior to enrolling the subject. If agreement is reached between the Investigator and Sponsor for the subject to continue in the study, all allowed medications should be maintained at a constant dose throughout the study.
4. The Principal Investigator deems any clinical laboratory test (at the Screening Visit) abnormality to be clinically significant
5. The subject has participated in other studies of investigational drugs or devices within 30 days prior to enrollment in this study (other than Study SPD426-406).
6. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
7. The subject has a concurrent chronic or acute illness, disability, or other condition (including significant unexpected laboratory or electrocardiogram [ECG] findings) that might confound the results of the tests and/or measurements administered in this study, or that might have increased the risk to the subject.
8. Known or suspected intolerance or hypersensitivity to the investigational product(s), closely-related compounds, or any of the stated ingredients.
9. Prior enrollment failure or randomization in this study.
10. History of alcohol abuse or other substance abuse within the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2013-06-22 (Actual); Study Completion 2013-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- United States (13):
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Advance Research Institute Inc, New Port Richey, Florida
  - Analab Clinical Research Inc, Lenexa, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Buffalo Clinical Research Center (BCRC), Buffalo, New York
  - NYU Medical Centre, New York, New York
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Kidney and Hypertension Center, Roseburg, Oregon
  - New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee
  - The Heartbeat Clinic, PA, McKinney, Texas
  - Aspen Clinical Research, Orem, Utah
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin

REFERENCES:
- [Result] Smith W, Wan H, Much D, Robinson AG, Martin P. Clinical benefit of midodrine hydrochloride in symptomatic orthostatic hypotension: a phase 4, double-blind, placebo-controlled, randomized, tilt-table study. Clin Auton Res. 2016 Aug;26(4):269-77. doi: 10.1007/s10286-016-0363-9. Epub 2016 Jul 2. PMID 27372462

RESULTS

PARTICIPANT FLOW:
Groups:
- Midodrine HCl (Open-label Phase): On the morning of Day -1, subjects took their usual morning dose of midodrine HCl, using their own midodrine HCl supplies at approximately the same time before rising that they would normally take their morning dose. On the morning of Day 1, subjects had their usual morning dose of midodrine HCl withheld.
- Placebo First, Then Midodrine HCl (Randomized Phase): Placebo for first intervention on Day 2, then Midodrine hydrochloride dose at the subject's current dose level for the second intervention on Day 3.
- Midodrine HCl First, Then Placebo (Randomized Phase): Midodrine hydrochloride dose at the subject's current dose level for the first intervention Day 2, then placebo for second intervention on Day 3.
Period: Open-label Phase
Arm/Group | Midodrine HCl (Open-label Phase) | Placebo First, Then Midodrine HCl (Randomized Phase) | Midodrine HCl First, Then Placebo (Randomized Phase)
Started | 24 | 0 | 0
Completed | 20 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Other | 4 | 0 | 0
Period: Randomized Phase (First Intervention)
Arm/Group | Midodrine HCl (Open-label Phase) | Placebo First, Then Midodrine HCl (Randomized Phase) | Midodrine HCl First, Then Placebo (Randomized Phase)
Started | 0 | 10 | 10
Completed | 0 | 9 | 10
Not Completed | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0
Period: Randomized Phase (Second Intervention)
Arm/Group | Midodrine HCl (Open-label Phase) | Placebo First, Then Midodrine HCl (Randomized Phase) | Midodrine HCl First, Then Placebo (Randomized Phase)
Started | 0 | 9 | 10
Completed | 0 | 9 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Safety Analysis Set defined as all subjects who received at least 1 dose of randomized investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Midodrine HCl (Randomized Phase) | Midodrine HCl First, Then Placebo (Randomized Phase) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (19.52) | 42.1 (18.64) | 45.1 (18.82)
Age, Customized [Count of Participants; unit: Participants]
  18 to 65 years, inclusive | 8 | 8 | 16
  >= 66 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Syncope/Near Syncope While on Tilt Table
Description: After a 30-minute supine period, the table was tilted from 0-90º within 30 seconds and maintained in that position for 45 minutes or until endpoint. Subjects were monitored for near-syncopal symptoms (subject felt sufficiently dizzy, lightheaded, faint, or felt like they were about to black out and requested the table to be returned to horizontal). Such a report ended the test. Alternatively, if the investigator observed that the subject was about to lose consciousness, that also constituted an endpoint.
Time Frame: 1 hour post-dose
Population: The Full Analysis Set was defined as all randomized subjects who received at least 1 dose of randomized investigational product and who had at least 1 measurement of the time to onset of syncopal symptoms/near syncope during tilt-table testing.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Midodrine HCl
Number analyzed (Participants) | 19 | 19
seconds | 1105.6 (186.82) | 1626.6 (186.82)
Statistical Analysis 1: Comparison: Placebo vs Midodrine HCl; Test type: Superiority or Other; p = 0.0131, ANOVA; Mean Difference (Final Values) = 521.0, 95% CI 2-sided [124.2 to 917.7]

ADVERSE EVENTS:
Groups:
- Midodrine HCl (Open-label Phase); Midodrine HCl (Randomized Phase): dose at the subject's current dose level
- Placebo (Randomized Phase): single dose of matching placebo
Arm/Group | Midodrine HCl (Open-label Phase) | Placebo (Randomized Phase) | Midodrine HCl (Randomized Phase)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/24 | 1/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midodrine HCl (Open-label Phase) (N=24) | Placebo (Randomized Phase) (N=20) | Midodrine HCl (Randomized Phase) (N=20)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.